CLINICAL TRIAL: NCT04976517
Title: A Multicenter Clinical Study of Echocardiographic Evaluation of the Impact of Diabetes and Prognostic Analysis of Heart Transplantation
Brief Title: Echocardiographic Assessment of the Impact of Diabetes and Prognostic Analysis of Heart Transplantation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xie Mingxing (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Shanghai Zhongshan Hospital (Other); Wuhan Asia Heart Hospital (Other); Guangdong Provincial People's Hospital (Other); Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Xie Mingxing, MD, PhD,FACC, FAHA, FASE, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Other Study IDs: 2021 v1.00
Record Dates: First submitted 2021-07-11; First posted 2021-07-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Heart Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- non-diabetes group: patients who underwent heart tranplantation without diabetes
- pre-transplant diabetes group: patients who underwent heart tranplantation with diabetes before the transplantation
- post transplant daibetes group: patients who underwent heart tranplantation without diabetes until after the transplantation

SUMMARY:
The aim of this study is to evaluat the impact of diabetes on cardiac function in patients with heart transplantation by multimodal imaging and analyse their prognosis.

DETAILED DESCRIPTION:
This study is planed to enroll 300000 patients after heart transplantation, all the patients will be divided into 3 groups according to whether or not they have diabetes and when did they develop diabete. Echocardiography will be used to evaluat their cardiac function. Comparing their cardiac function and clinical information and analysing their prognosis to evaluat the impact of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who received a heart transplant after 2015

Exclusion Criteria:

* The image quality is poor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who received a heart transplant after 2015
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | up to 2023.12
  death from all causes
acute rejection | up to 2023.12
  acute rejection required treatment
readmission | up to 2023.12
  readmission from all causes

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, PhD, Principal Investigator — Department of Ultrasound, Union Hospital, Wuhan, China

IPD SHARING:
Plan to Share IPD: No